CLINICAL TRIAL: NCT00773149
Title: Phase I/II Study of Alemtuzumab (CAMPATH 1H) Associated to G-CSF in Adult Patients With Refractory Acute Lymphocytic Leukemia (ALL) or ALL in Relapse.
Brief Title: Alemtuzumab (CAMPATH 1H) Associated to G-CSF in Adult Patients With Refractory Acute Lymphocytic Leukemia
Acronym: Campath
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P051003
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2011-02

CONDITIONS: Acute Lymphocytic Leukemia
Keywords: Adult Acute Lymphocytic Leukemia; Alemtuzumab
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): all included patients
  Interventions: Drug: Alemtuzumab (CAMPATH 1H) associated to G-CSF

INTERVENTIONS:
Drug: Alemtuzumab (CAMPATH 1H) associated to G-CSF — All patients receive Alemtuzumab in 3 successive phases:
  Phase A: Test week: 3mg, then 10mg, then 30mg every other day for one week to test for tolerance.
  Phase B: 30mg 3 times a week for 12 to 18 administrations until response or progression/failure has been documented.
  Phase C: in patients in CR, maintenance with Alemtuzumab: 3 injections one week every 2 months.

SUMMARY:
Alemtuzumab is an anti CD52 monoclonal antibody. The CD52 antigen is present at the surface of B,T NK lymphocytes. It is expressed at various levels at the surface of ALL blast cells. Adult patients with ALL in relapse have less than 10% probability of long term survival. The present study will test the response rate (partial and complete remission) of refractory ALL or ALL in relapse. It is hoped that if a CR can be achieved, further consideration will be given for a hematopoietic stem cell transplant.

The use of G-CSF is justified by a possible increase in ADCC.

DETAILED DESCRIPTION:
All patients receive Alemtuzumab in 3 successive phases:

Phase A: Test week: 3mg, then 10mg, then 30mg every other day for one week to test for tolerance.

Phase B: 30mg 3 times a week for 12 to 18 administrations until response or progression/failure has been documented.

Phase C: in patients in CR, maintenance with Alemtuzumab: 3 injections one week every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 15 years
* Refractory ALL
* ALL in relapse post chemotherapy or post transplant
* ALL blast cells expressing CD 52 antigen at any time during the evolution of the disease.
* Signed informed consent
* Patients under social security coverage
* Anti conceptional tablets in pre menopausal women.

Exclusion Criteria:

* Children below 15 years of age or aged 15
* Blast cells not expressing CD52 antigen (at all evaluations)
* HIV positivity
* ECOG Score 3 and 4
* Hypersensitivity to Alemtuzumab.
* Pregnancy or breast feeding.
* Other malignant disease in addition to ALL.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-10; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Partial and complete remission, overall response rates | At 2 years

SECONDARY OUTCOMES:
Valuation of tolerance, more particularly targeted at the immunodeficiency shortage, contagious complications and neurotoxicity assessed according to the NCI (National Cancer Institute) classification. | At 2 years
Valuation of the response waiting time, from the first day of the induction treatment to the REEVOLUTING. | at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Claude GORIN, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Saint Antoine Hospital, Hematology Unit, Paris, France